CLINICAL TRIAL: NCT03480867
Title: Pre-operative Radiation Therapy (RT) and Temozolomide (TMZ) in Patients With Newly Diagnosed Glioblastoma. A Phase I Study. (PARADIGMA)
Brief Title: Pre-operative RT and TMZ in Patients With Newly Diagnosed GBM Diagnosed Glioblastoma. A Phase I Study. (PARADIGMA)
Acronym: PARADIGMA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: competing study was opened by the surgeon after this trial was opened
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Valerie Panet-Raymond, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUHC-2016-1524
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Glioblastoma Multiforme, Adult
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: RT 28Gy in 7 fractions with a concomitant boost of 42Gy in 7 fractions+ Temozolomide (75mg/m2) followed by surgery then Temozolomide (150-200mg/m2) q 5 days every 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-operative RT and TMZ (Experimental): * Single Arm: Pre-operative Radiation +Temozolomide followed by Surgery plus six cycles of Temozolomide
  Interventions: Drug: Temozolomide; Radiation: Pre-Operative Radiation

INTERVENTIONS:
Drug: Temozolomide — Experimental: Registered one arm study Seven days of pre-operative Radiation+Temozolomide followed by surgery plus TMZ, as adjuvant component.for six cycles.
  Other Names: Surgery
Radiation: Pre-Operative Radiation — Radiation is given with Temozolomide for 7 days before surgery

SUMMARY:
Glioblastoma (GBM) is the most common primary brain cancer in adults. Despite surgery, conventional radiotherapy, and chemotherapy, the average survival for GBM is 15-16 months. Although additional chemoradiotherapy has been shown to increase survival, the majority recur at the original location.

Despite many efforts to improve the local control by improving surgical techniques, increasing the radiotherapy dose or adding newer chemotherapy agents, these attempts have failed to show a survival benefit or an improved cancer control. People who are not participating in a study are usually treated with surgery followed by radiation (6 weeks duration) together with temozolomide (chemotherapy drug) followed by temozolomide alone. For patients who receive this usual treatment approach for this cancer, about 4 out of 100 are free of cancer growth five years later. Because GBM invades the surrounding normal brain, this study is looking into the possibility of minimizing invasion by starting treatment using the combination of radiotherapy and chemotherapy prior to surgery. This approach is an experimental form of treatment and the diagnosis is based exclusively on imaging and not on histology of the tumour tissue, and there is a possibility that your tumor may not be a GB but of other origins.

DETAILED DESCRIPTION:
One of the deadly properties of GBM is its capacity to diffusely infiltrate the surrounding normal brain tissue. Unlikely many malignancies, in GBM local disease progression, rather than metastatic disease, is the leading cause of death. Extent of resection plays a key role in the treatment of these patients with complete surgical resection improving outcome. In a prospective, non- interventional, multi-institutional study of over 140 patients with GBM and minimal or no residual tumor on post-operative MRI, Stummer et al.have shown that extent of resection is indeed associated with improved survival. However, despite evidence of complete resection on post-operative imaging studies, surgery is rarely truly complete. GBMs are invasive tumors and, at time of surgery, a clear boundary is not clearly identifiable, either on pre- or intra- operative imaging. Even when sophisticated imaging'techniques are used, they are unable to detect invasive brain cancer cell for proper pre-operative surgical planning to optimally delineate the tumor boundaries for a truly complete resection. Even if they were, brain eloquence would preclude a complete resection of most GBMs.

Despite extensive and complete surgical tumor removal coupled with radiation and chemotherapy, even in high doses, 90% of patients still fail at the border or within a few centimeters from the surgical cavity. Glioma cell migration outside the original tumor site may be responsible for this recurrence pattern. Cell migration is a complex, dynamic process and is well-documented in GBM. It involves, at least, 3 independent but coordinated biologic processes: 1) cell adhesion to components of the extracellular matrix, 2) cell's own motility and 3) invasion. Giese et al.) reported that cell migration is established by several independent mechanisms, facilitating the spread of tumor astrocytes, but with cell motility being the possible common denominator for this biologic behavior.

Invasion of tumor glioma cells is a multi-factorial process. To migrate, the cell needs a change in morphology and to interact with the extracellular matrix. It is possible that the surgical insult at the time of tumor removal may facilitate such an environment. Also, Wild-Bode et al.(6) have shown, in animal models, that sub-lethal doses of irradiation promote the migration and invasiveness of glioma cells. It is conceivable that the use of conventionally fractionated radiation therapy (2 Gy per day), even in doses above 60 Gy, leads to only sub-lethal damage potentially promoting cell migration.

In a recently completed Phase 2 study for patients with newly diagnosed GBM, our group has shown that the use of concurrent temozolomide and hypofractionated radiation therapy to a dose of 60 Gy given in 20 fractions (daily dose of 3 Gy) preceded by 2 weeks of temozolomide given in the post-operative setting was associated with 2-year survival rates of 63% and 29% for MGMT methylated and unmethylated tumors, respectively (Dr. G. Shenouda, personal information. Manuscript submitted for publication). These promising results may be possibly due to a dual effect of the use of neoadjuvant temozolomide (prior to radiation therapy) and the use of a hypofractionated radiotherapy regimen. The upfront use of temozolomide may have affected tumor control by interfering with the upstream signaling event triggered by the RT preventing cell migration and also by promoting inhibition of glioma cell invasion.

GBMs are one of the most rapidly growing tumors. Primary GBMs typically develop and grow to be greater than 3 cm in less than 4 months. Under the current standard treatment approach, patients undergo surgery and, rather than starting adjuvant therapy immediately at a moment when there is the least amount of residual tumor burden, they wait 3-4 weeks, for practical reasons, to start adjuvant treatment with RT and TMZ. In addition, the combined treatment takes an additional 6 weeks to complete. Thus it takes 9-10 weeks for patients to complete maximum local treatment. In other words, one of the most aggressive tumors has been given another 9-10 weeks to proliferate, repopulate and invade. It is conceivable that this delay in adjuvant treatment gives the residual brain cancer cells the opportunity to regrow and invade prior to completion of RT and TMZ thus contributing to 85% of all failures occurring at or within 2 cm of the original resection cavity margin.

The use of pre-operative RT, either alone or in combination with chemotherapy, has been successfully used in other pathologies. In patients with soft tissue sarcoma, localized . rectal cancer, locally advanced breast cancer, and esophageal cancer the use of pre-operative RT has been associated with improved local control (8-11). Recently, the use of neoadjuvant radiosurgery has been explored in patients harboring resectable metastatic brain lesions (12). A total of 47 patients underwent radiosurgery prior to the surgical procedure (total of 51 lesions) and the authors report high rates of local control with limited toxicity. The use of pre-operative RT has several theoretical advantages in patients with GBM. Neoadjuvant RT is delivered prior to the surgical procedure minimizing, theoretically, the risk of local cell migration at the time of the surgical intervention. It has also the advantage of treating a target that has an intact blood supply and, most importantly, RT will be delivered to a better defined target. It also allows a definitive portion of the treatment paradigm to be delivered in a timely manner with no prolonged delay.

ELIGIBILITY:
Inclusion Criteria

* Newly diagnosed (MR image-based) GBM - Must be able to undergo gadolinium-enhanced MRI.
* Must be a candidate for radical surgical resection in the opinion of the neurosurgeon.
* The tumor must measure less than 6 cm in maximum diameter. The tumor diameter will be the greatest diameter as measured on the contrast-enhanced MRI.
* A neurosurgical oncologist, radiation oncologist and neuro-oncologist will assess each patient in advance of enrollment.
* The estimated post-surgical radiation field must be compatible with the proposed radiation scheme - ie, to ensure a safe radiation margin from structures such as the optic apparatus and brain stem.
* The GBM tumor must be located in the supratentorial compartment only (any component involving the brain stem or cerebellum is not allowed)
* Age>18years
* Karnofsky Performance Status (KPS) 70.
* History and physical examination within 14 days from start of therapy, including documentation of steroid dose.
* Adequate complete blood counts (Absolute neutrophil count (ANC) .:! 1,800. cells/mm3; Platelets.:! 100,000 cells/mm3; Hemoglobin.:! 10.0 g/dl), renal and liver function within 14 days prior to therapy with values< 3x (upper limit normal) ULN.
* For females of child-bearing potential, negative serum pregnancy test within 14 days prior to therapy and use of contraception.
* Signed consent form.

Exclusion Criteria:

* Tumors within 1 cm from critical structures (brainstem, optic apparatus), or with massive edema, or with the possibility of herniation, or any tumor that in the neurosurgeon's opinion would be considered unsafe to delay surgery or is not grossly resectable.
* Prior invasive malignancy (except for non-melanomatous skin cancer, non- invasive bladder cancer, and non-invasive cervix cancer) unless disease free for 2:5 years.
* Recurrent or multifocal GBM.
* Any site of metastatic disease (drop metastases).
* Prior chemotherapy or radiation therapy to the head or neck (except for T1 glottic tumor
* Severe active co-morbid medical condition as assessed by medical team.
* Patients enrolled in any other protocol.
* Inability to undergo MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
To assess toxicity of the regimen | one year
  Toxicity will be assessed and graded using CTCAE V. 4.03

SECONDARY OUTCOMES:
Number of patients completing the study treatment | one year.
  To determine the overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Panet-Raymond, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre-Cedars Cancer Centre, Montreal, Québec, Canada, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Upon official request approved by the Research Ethics Board (REB), some data may be shared depending on what needs to be shared.

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Gilbert MR, Dignam JJ, Armstrong TS, Wefel JS, Blumenthal DT, Vogelbaum MA, Colman H, Chakravarti A, Pugh S, Won M, Jeraj R, Brown PD, Jaeckle KA, Schiff D, Stieber VW, Brachman DG, Werner-Wasik M, Tremont-Lukats IW, Sulman EP, Aldape KD, Curran WJ Jr, Mehta MP. A randomized trial of bevacizumab for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):699-708. doi: 10.1056/NEJMoa1308573. PMID 24552317
- [Background] Stummer W, Meinel T, Ewelt C, Martus P, Jakobs O, Felsberg J, Reifenberger G. Prospective cohort study of radiotherapy with concomitant and adjuvant temozolomide chemotherapy for glioblastoma patients with no or minimal residual enhancing tumor load after surgery. J Neurooncol. 2012 May;108(1):89-97. doi: 10.1007/s11060-012-0798-3. Epub 2012 Feb 4. PMID 22307805
- [Background] Giese A, Bjerkvig R, Berens ME, Westphal M. Cost of migration: invasion of malignant gliomas and implications for treatment. J Clin Oncol. 2003 Apr 15;21(8):1624-36. doi: 10.1200/JCO.2003.05.063. PMID 12697889
- [Background] Wild-Bode C, Weller M, Rimner A, Dichgans J, Wick W. Sublethal irradiation promotes migration and invasiveness of glioma cells: implications for radiotherapy of human glioblastoma. Cancer Res. 2001 Mar 15;61(6):2744-50. PMID 11289157
- [Background] Wick W, Wick A, Schulz JB, Dichgans J, Rodemann HP, Weller M. Prevention of irradiation-induced glioma cell invasion by temozolomide involves caspase 3 activity and cleavage of focal adhesion kinase. Cancer Res. 2002 Mar 15;62(6):1915-9. PMID 11912174
- [Background] O'Sullivan B, Davis AM, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Kandel R, Goddard K, Sadura A, Pater J, Zee B. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet. 2002 Jun 29;359(9325):2235-41. doi: 10.1016/S0140-6736(02)09292-9. PMID 12103287
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Urschel JD, Vasan H. A meta-analysis of randomized controlled trials that compared neoadjuvant chemoradiation and surgery to surgery alone for resectable esophageal cancer. Am J Surg. 2003 Jun;185(6):538-43. doi: 10.1016/s0002-9610(03)00066-7. PMID 12781882
- [Background] Matuschek C, Bolke E, Roth SL, Orth K, Lang I, Bojar H, Janni JW, Audretsch W, Nestle-Kraemling C, Lammering G, Speer V, Gripp S, Gerber PA, Buhren BA, Sauer R, Peiper M, Schauer M, Dommach M, Struse-Soll K, Budach W. Long-term outcome after neoadjuvant radiochemotherapy in locally advanced noninflammatory breast cancer and predictive factors for a pathologic complete remission : results of a multivariate analysis. Strahlenther Onkol. 2012 Sep;188(9):777-81. doi: 10.1007/s00066-012-0162-8. Epub 2012 Aug 11. PMID 22878547
- [Background] Asher AL, Burri SH, Wiggins WF, Kelly RP, Boltes MO, Mehrlich M, Norton HJ, Fraser RW. A new treatment paradigm: neoadjuvant radiosurgery before surgical resection of brain metastases with analysis of local tumor recurrence. Int J Radiat Oncol Biol Phys. 2014 Mar 15;88(4):899-906. doi: 10.1016/j.ijrobp.2013.12.013. PMID 24606851
- [Background] Law M, Yang S, Wang H, Babb JS, Johnson G, Cha S, Knopp EA, Zagzag D. Glioma grading: sensitivity, specificity, and predictive values of perfusion MR imaging and proton MR spectroscopic imaging compared with conventional MR imaging. AJNR Am J Neuroradiol. 2003 Nov-Dec;24(10):1989-98. PMID 14625221
- [Background] Warren KE, Patronas N, Aikin AA, Albert PS, Balis FM. Comparison of one-, two-, and three-dimensional measurements of childhood brain tumors. J Natl Cancer Inst. 2001 Sep 19;93(18):1401-5. doi: 10.1093/jnci/93.18.1401. PMID 11562391
- [Background] Boxerman JL, Ellingson BM, Jeyapalan S, Elinzano H, Harris RJ, Rogg JM, Pope WB, Safran H. Longitudinal DSC-MRI for Distinguishing Tumor Recurrence From Pseudoprogression in Patients With a High-grade Glioma. Am J Clin Oncol. 2017 Jun;40(3):228-234. doi: 10.1097/COC.0000000000000156. PMID 25436828
- [Background] Mangla R, Singh G, Ziegelitz D, Milano MT, Korones DN, Zhong J, Ekholm SE. Changes in relative cerebral blood volume 1 month after radiation-temozolomide therapy can help predict overall survival in patients with glioblastoma. Radiology. 2010 Aug;256(2):575-84. doi: 10.1148/radiol.10091440. Epub 2010 Jun 7. PMID 20529987
- [Background] Law M, Young RJ, Babb JS, Peccerelli N, Chheang S, Gruber ML, Miller DC, Golfinos JG, Zagzag D, Johnson G. Gliomas: predicting time to progression or survival with cerebral blood volume measurements at dynamic susceptibility-weighted contrast-enhanced perfusion MR imaging. Radiology. 2008 May;247(2):490-8. doi: 10.1148/radiol.2472070898. Epub 2008 Mar 18. PMID 18349315
- [Background] Cao Y, Tsien CI, Nagesh V, Junck L, Ten Haken R, Ross BD, Chenevert TL, Lawrence TS. Survival prediction in high-grade gliomas by MRI perfusion before and during early stage of RT [corrected]. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):876-85. doi: 10.1016/j.ijrobp.2005.09.001. Epub 2005 Nov 18. PMID 16298499
- [Background] Costa BM, Smith JS, Chen Y, Chen J, Phillips HS, Aldape KD, Zardo G, Nigro J, James CD, Fridlyand J, Reis RM, Costello JF. Reversing HOXA9 oncogene activation by PI3K inhibition: epigenetic mechanism and prognostic significance in human glioblastoma. Cancer Res. 2010 Jan 15;70(2):453-62. doi: 10.1158/0008-5472.CAN-09-2189. Epub 2010 Jan 12. PMID 20068170
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676